CLINICAL TRIAL: NCT00695864
Title: Effect of Ondansetron for Withdrawal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Principle Investigator, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SU-05222008-1180; 14228
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Substance Withdrawal Syndrome
MeSH Terms: conditions — Substance Withdrawal Syndrome | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Placebo - sugar pill (Placebo Comparator): Placebo - sugar pill
  Interventions: Drug: Ondansetron and Placebo crossover
- Ondansetron (Experimental): Ondansetron
  Interventions: Drug: Ondansetron and Placebo crossover

INTERVENTIONS:
Drug: Ondansetron and Placebo crossover

SUMMARY:
We hope to determine whether Ondansetron, an anti-nausea medication, works to help relieve withdrawal symptoms experienced while the patient is being weaned off opioid medications. This medication has shown anecdotal evidence of being affective for the treatment of withdrawal symptoms and we hope to determine whether this is affective.

ELIGIBILITY:
Inclusion Criteria:-Over 18 years of age

* No medical contraindications to medication
* Able to fulfill research procedures Exclusion Criteria:-Subjects who are unable to respond to our questionnaires or to stimuli as required by the experimental protocol will be excluded.
* Subjects will be excluded if they have a history of significant psychiatric disorders that would prevent them from engaging in a treatment program.
* Participating in other studies that would interfere with the procedures in this study
* Known or apparent pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Mackey, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 31 patients enrolled, 17 did not experience withdrawal symptoms and were therefore not assigned an intervention.
Groups:
- Placebo Then Ondansetron: Dosage and form:
  Placebo - tablet Odansetron - 8 mg oral tablet
  Double-blind, placebo-controlled, cross-over trial. All participants received placebo first, followed by Ondansetron.
Period: Placebo
Arm/Group | Placebo Then Ondansetron
Started | 14
Completed | 9
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 4
Period: Ondansetron
Arm/Group | Placebo Then Ondansetron
Started | 14
Completed | 9
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Placebo Then Ondansetron
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 42.8 [27 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Withdrawal Symptoms With Placebo and With Ondansetron
Description: Subjective Opioid Withdrawal Scale: Participants were asked to rate, from 0 to 4, their experience of 15 withdrawal symptoms. Scores for each participant were derived from the sum of their withdrawal symptoms score (minimum:0, maximum: 60). A higher score indicates more symptoms experienced and/or at a greater degree of severity.
Time Frame: Baseline, 1 hour post dose Placebo, 1 hour post dose Ondansetron
Population: 9 participants and 13 independent trials (3 patients had more than 1 distinct withdrawal episode) were analyzed. Of the 14 participants assigned to intervention, 5 were withdrawn from the study and/or analysis.
Measure: Mean (Standard Error); unit: Percent change
Groups:
- Placebo - Sugar Pill: Placebo - sugar pill
  Ondansetron and Placebo crossover
- Ondansetron: Ondansetron
  Ondansetron and Placebo crossover
Arm/Group | Placebo - Sugar Pill | Ondansetron
Number analyzed (Participants) | 9 | 9
Percent change | -22.08 (8.61) | -42.71 (7.47)

ADVERSE EVENTS:
Arm/Group | Placebo - Sugar Pill | Ondansetron
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes